CLINICAL TRIAL: NCT00064675
Title: Genetics of Cardiovascular Reactivity in Black Youth
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1229; R01HL072375 (NIH); R01HL068971-04 (NIH)
Record Dates: First submitted 2003-07-10; First posted 2003-07-14 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — buccal specimens stored at Med Coll Wisconsin

SUMMARY:
To evaluate individual differences in cardiovascular responses to acute stress in Black adolescents.

DETAILED DESCRIPTION:
BACKGROUND:

The prevalence and severity of essential hypertension (EH) are greater among Black Americans than other ethnic groups in the U.S. Blacks are at increased risk for target organ damage from elevated blood pressure, including heart disease, stroke, and endstage renal failure. There are significant ethnic differences in cardiovascular reactivity (CVR) to stress, which is a risk factor for elevated blood pressure. Studies have shown that CVR to stress is stable over time, heritable, and predictive of future elevations in blood pressure and the development of essential hypertension. These properties make measures of CVR a valuable intermediate for genetic studies of hypertensive risk.

DESIGN NARRATIVE:

The genetic epidemiology study will test the hypothesis that individual differences in CVR to acute stress in Black youth are associated with well defined polymorphisms in candidate genes related to blood pressure including: 1) alpha- and beta-adrenergic receptor genes; 2) genes involved in catecholamine metabolism; 3) genes involved in endocrine function; 4) genes involved in the renin angiotensin system. By focusing on normotensive youth at risk for developing essential hypertension, the investigators hope to identify genes associated with the onset, rather than the sequelae, of hypertension. Moreover, given that CVR to acute stress is defined as a change in cardiovascular function evoked by an environmental manipulation of stress, the research is inherently a study of gene-environment interactions.

A total of 500 unrelated Black adolescents and young adults (equal numbers of males and females), 15-21 years of age will be studied. Buccal cell samples will be collected for DNA extraction from all subjects for genetic association analyses. Impedance cardiography and blood pressure monitoring will be used to assess components of CVR to stress during video game, mental arithmetic, cold pressor, and whole body cold exposure tasks, all of which have been utilized or developed in the laboratory. Various methods will be used to evaluate genetic associations with CVR to acute stress, including analyses of single nucleotide polymorphisms and haplotypes. Supplementary analyses will evaluate potential gene-gene interactions and additional gene-environment interactions involving chronic environmental stress.

ELIGIBILITY:
African American non-hypertensive, no chronic disease which would affect blood pressure

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 500 African American youth
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
genes associated with hyperreactivity | done
  several genes associated with reactivity

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Alpert, Principal Investigator — University of Tennessee